CLINICAL TRIAL: NCT01303237
Title: A Post Marketing Surveillance Study to Assess the Safety and Efficacy of Cetuximab Plus Radiotherapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck (LA SCCHN)
Brief Title: A Post Marketing Surveillance Study to Assess the Safety and Efficacy of Cetuximab Plus Radiotherapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Acronym: PMS LAD SCCHN
Status: Terminated | Type: Observational
Why Stopped: The study was discontinued due to slow recruitment and subjects not completing follow up period.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd., India (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR062202-539
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Unresectable Locally Advanced Squamous Cell Carcinoma of Head and Neck; LA SCCHN
Keywords: LA SCCHN; Cetuximab; RT; PMS
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab + RT — Cetuximab initial dose 400 mg/m² on week 1; Cetuximab maintenance dose 250 mg/m² continued for 7 weeks plus concomitant RT
  Other Names: Erbitux

SUMMARY:
This prospective, observational, multicentre, post marketing surveillance study will collect safety and efficacy information on patients with Locally Advanced Squamous Cell Carcinoma of the Head and Neck (LA SCCHN) treated with Cetuximab and Radiotherapy (RT) based on the locally approved label.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, observational, single arm, cohort study, wherein 200 patients of unresectable LA SCCHN will be enrolled. The eligibility of the patients will be decided by the Investigators based on the locally approved label. The patients will be treated with Cetuximab in combination with RT for a duration of 8 weeks and then followed up for 3 years. The objectives of this study are to record safety and efficacy information on the treatment combination in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria as per the product label for LA SCCHN approved by India Health Authority
* Unresectable Locally Advanced Squamous Cell Carcinoma of the Head and Neck
* Patient willing and able to give written Informed Consent
* Patient capable of complying with study data collection procedures

Exclusion Criteria:

* Exclusion criteria as per the product label for LA SCCHN approved by India Health Authority

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unresectable Locally Advanced (Stage III/ IV A or IV B) SCCHN patients found eligible to receive Cetuximab + RT
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-02-28 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2014-08-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Serious Adverse Reactions | 3 years
  Number of patients with Serious Adverse Reactions will be assessed to discover the tolerability of the treatment regimen.

SECONDARY OUTCOMES:
Response Rate | 3 years
Progression Free Survival | 3 years
Duration of Locoregional Disease Control | 3 years
Overall Survival | 3 years
Response Rate | 8 weeks (Post completion of treatment duration)
Management of skin conditions due to treatment protocol | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Rana, MD, Study Director — Merck Ltd., India
Locations (25):
- India (25):
  - Omega Hospital, Hyderabad, Andhra Pradesh
  - Shanti Chandra Family Clinic, Hyderabad, Andhra Pradesh
  - Swarna Sai Hospital, Hyderabad, Andhra Pradesh
  - Dr. Nikhil's Clinic, Secunderabad, Andhra Pradesh
  - Arogya Multispeciality Clinic, Mangalore, Bangalore
  - Aastha Oncology Associates, Ahmedabad, Gujarat
  - Navneet Memorial Centre, Ahmedabad, Gujarat
  - Meharbai TATA Memorial Hospital, Bistupur, Jamshedpur
  - Dr. T. P. Sahoo's Clinic, Bhopal, Madhya Pradesh
  - Ruby Hall Clinic, Pune, Maharashtra
  - Dr S M Karandikar Hospital, Pune, Maharashtra
  - Dwidal Nursing Home, Pune, Maharashtra
  - Regional cancer center, Sheikpura, Patna
  - Grecian Superspeciality Hospital, Mohali, Punjab
  - Harmony Health Care, Mohali, Punjab
  - Bhagwan Mahaveer Cancer Hospital & Research Center, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Cancer Care Centre, Jaipur, Rajasthan
  - Balaji Clinic & General Hospital, Jaipur, Rajasthan
  - Royal Cancer Institute and Research Centre, Kanpur, Uttar Pradesh
  - SMH Curie Cancer Centre, New Delhi, Uttar Pradesh
  - Bengal Oncology, Kolkata, West Bengal
  - Apollo Gleneagles Cancer Hospital, Kolkata, West Bengal
  - Oncologist & Palliative Care Specialist Clinic, Kolkata, West Bengal
  - Dr. Meenu's Clinic, Delhi